CLINICAL TRIAL: NCT02081274
Title: Influence of Tidal Volume During Mechanical Ventilation on Postoperative Clinical Outcome in Pediatric Patients Undergoing Congenital Heart Surgery
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, WonHo Kim, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-12-146
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Patients Who Underwent Surgery for Congenital Heart Disease
Keywords: tidal volume; congenital heart disease; mortality
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients who underwent surgery for congenital heart disease: patients who underwent surgery for congenital heart disease between 2009 and 2013 in Samsung Medical Center
  Interventions: Procedure: Surgery for congenital heart disease

INTERVENTIONS:
Procedure: Surgery for congenital heart disease

SUMMARY:
High tidal volume during mechanical ventilation has been reported to increase mortality in patients with acute lung injury or acute respiratory distress syndrome. High tidal volume was also reported to be associated with increased mortality in adult patients without acute lung injury or acute respiratory distress syndrome. However, the influence of high tidal volume on clinical outcome in pediatric patients who underwent surgery for congenital heart disease has not been evaluated yet. The investigators attempted to evaluate the effect of tidal volume on clinical outcome in both cyanotic and non-cyanotic congenital heart disease.

DETAILED DESCRIPTION:
High tidal volume during mechanical ventilation has been reported to increase mortality in patients with acute lung injury or acute respiratory distress syndrome. High tidal volume was also reported to be associated with increased mortality in adult patients without acute lung injury or acute respiratory distress syndrome. However, the influence of high tidal volume on clinical outcome in pediatric patients who underwent surgery for congenital heart disease has not been evaluated yet. The investigators attempted to evaluate the effect of tidal volume on clinical outcome in both cyanotic and non-cyanotic congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients who underwent surgery for congenital heart disease with cardiopulmonary bypass between 2009 and 2013 in Samsung Medical Center

Exclusion Criteria:

* patients who lack data regarding mortality, creatinine, estimated glomerular filtration rate, or urine output.

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric patients who underwent surgery for congenital heart disease with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient Mortality | six month after surgery
  Patient Mortality at six month after surgery

SECONDARY OUTCOMES:
Patient Mortality | in-hospital, one-month, and one-year after surgery
  In-hospital, one-month and one-year mortality after surgery
acute kidney injury as defined by RIFLE criteria (for Risk, Injury, Failure, Loss, End-stage kidney disease) | during one week after surgery
  acute kidney injury as defined by RIFLE criteria (for Risk, Injury, Failure, Loss, End-stage kidney disease)

CONTACTS AND LOCATIONS:
Overall Officials: Won Ho Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea